CLINICAL TRIAL: NCT00098943
Title: Phase I Trial of NGR-TNF Administered Every 3 Weeks as a 1 Hour Intravenous Infusion in Patients With Solid Tumor
Brief Title: NGR-TNF in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16041; EORTC-16041; MOLMED-EORTC-16041; EUDRACT-2004-000950-21
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer; Head and Neck Cancer; Kidney Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage IV renal cell cancer; recurrent renal cell cancer; stage IV colon cancer; recurrent colon cancer; anaplastic thyroid cancer; insular thyroid cancer; thyroid gland medullary carcinoma; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer; recurrent thyroid cancer; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent verrucous carcinoma of the larynx; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; metastatic parathyroid cancer; recurrent parathyroid cancer; recurrent salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell; Colonic Neoplasms; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Parathyroid Neoplasms; Salivary Gland Neoplasms | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

INTERVENTIONS:
Biological: CNGRC peptide-TNF alpha conjugate

SUMMARY:
RATIONALE: Targeted therapy with tumor necrosis factor combined with a fusion protein may stop the growth of solid tumors by stopping blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of NGR-TNF in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of tumor vasculature-targeted tumor necrosis factor alpha (NGR-TNF) in patients with advanced solid tumors.
* Determine the recommended phase II dose of this drug in these patients.

Secondary

* Determine the mechanism of action of this drug in these patients.
* Determine response in patients treated with this drug.

OUTLINE: This is an open-label, nonrandomized, dose-escalation, multicenter study.

Patients receive tumor vasculature-targeted tumor necrosis factor alpha (NGR-TNF) IV over 1 hour on day 1. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 1-6 patients receive escalating doses of NGR-TNF until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients receive treatment at the MTD.

Patients are followed every 8 weeks until disease progression or the start of a new anticancer treatment.

PROJECTED ACCRUAL: A total of 1-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced solid tumor not amenable to any clinical improvement by current standard treatments

  * Preferably tumors well known to be very angiogenic (e.g., renal, colon, thyroid, and head and neck cancers)
* No clinical signs of CNS involvement

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2 OR
* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and/or ALT < 2.5 times ULN (5 times ULN in the presence of liver metastases)

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* Cardiac function normal
* No uncontrolled hypertension
* No condition in which hypovolemia and its consequences (e.g., increased stroke volume, elevated blood pressure) or hemodilution could represent a risk to the patient

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active or uncontrolled systemic infection
* No other uncontrolled disease, serious illness, or medical condition that would preclude study participation
* No known hypersensitivity/allergic reaction to human albumin preparations or any of the excipients
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 28 days since prior immunotherapy

Chemotherapy

* At least 28 days since prior chemotherapy and recovered

Endocrine therapy

* At least 28 days since prior hormonal therapy

Radiotherapy

* At least 28 days since prior radiotherapy and recovered
* No prior radiotherapy to > 25% of bone marrow reserve

Surgery

* More than 2 weeks since prior surgery

Other

* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose as measured by CTC v 3.0

SECONDARY OUTCOMES:
Clinical response as measured by RECIST criteria
Mechanism of action as measured by Dynamic Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J. A. Punt, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (2):
- University Medical Center Hamburg - Eppendorf, Hamburg, Germany
- Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Result] van Laarhoven HW, Fiedler W, Desar IM, van Asten JJ, Marreaud S, Lacombe D, Govaerts AS, Bogaerts J, Lasch P, Timmer-Bonte JN, Lambiase A, Bordignon C, Punt CJ, Heerschap A, van Herpen CM. Phase I clinical and magnetic resonance imaging study of the vascular agent NGR-hTNF in patients with advanced cancers (European Organization for Research and Treatment of Cancer Study 16041). Clin Cancer Res. 2010 Feb 15;16(4):1315-23. doi: 10.1158/1078-0432.CCR-09-1621. Epub 2010 Feb 9. PMID 20145168
- [Result] Van Laarhoven H, Fiedler W, Desar IM, et al.: Phase I and DCE-MRI evaluation of NGR-TNF, a novel vascular targeting agent, in patients with solid tumors (EORTC 16041). [Abstract] J Clin Oncol 26 (Suppl 15): A-3521, 2008.
- [Result] Heerschap A, Fiedler W, Marreaud S, et al.: A phase I study of NGR-TNF, a novel vascular targeting agent, in patients with refractory solid tumors (EORTC 16041). [Abstract] J Clin Oncol 25 (Suppl 18): A-14074, 2007.
- [Result] van Herpen C, Fiedler W, Marreaud S, et al.: A biological and pharmacologic phase I study of NGR-TNF, a novel vascular targeting agent, in patients with refractory solid tumors (EORTC 16041). [Abstract] American Association for Cancer Research: Molecular Targets and Cancer Therapeutics, October 22-26, 2007, San Francisco, CA A-B78, 2007.
- [Result] van Herpen C, Fiedler W, Toma S, et al.: Phase I study of NGR-TNF, a novel vascular targeting agent, in patients with refractory solid tumours (EORTC 16041). [Abstract] European Journal of Cancer Supplements 4 (12): A-366, 113, 2006.